CLINICAL TRIAL: NCT00406497
Title: Phase 2a Study of 0.05% Difluprednate Ophthalmic Emulsion in the Treatment of Postoperative Inflammation
Brief Title: Study of Difluprednate Ophthalmic Emulsion in the Treatment of Postoperative Inflammation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SJE2079/2-03-PC
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation

INTERVENTIONS:
Drug: Difluprednate Ophthalmic Emulsion

SUMMARY:
The purpose of this phase 2 study is to determine if difluprednate ophthalmic emulsion is effective in the treatment of postoperative inflammation.

DETAILED DESCRIPTION:
The objective is to assess efficacy endpoints in comparison with 0.1% BM ophthalmic solution, prior to investigation of the efficacy and safety of 0.05% DFBA ophthalmic emulsion in the treatment of postoperative intraocular inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing intraocular surgery (cataract surgery, cataract surgery + implantation of intraocular lens, vitreous surgery, cataract surgery + implantation of intraocular lens + vitreous surgery)
* Patients with anterior chamber cell score ≥2 on the next day of surgery
* Male and female patients aged ≥20 years (on the day of obtaining informed consent)
* Patients giving written informed consent prior to initiation of the study

Exclusion Criteria:

* Patients who did not meet all of the above inclusion criteria
* Patients receiving systemic administration of any corticosteroid or immunosuppressive drug, or topical application of corticosteroid ophthalmic ointment within 1 week before instillation of the investigational product
* Patients receiving topical injection of any corticosteroid in eyes before instillation of the investigational product (aqueous preparation: within 1 week before instillation of the investigational product, depot preparation: within 2 weeks before instillation of the investigational product)
* Patients receiving systemic administration of any non-steroidal anti-inflammatory drug or antiphlogistic enzyme
* Patients receiving instillation of any corticosteroid, non-steroidal anti-inflammatory ophthalmic solution or antiphologistic enzyme within 24 hours before ophthalmic examination prior to instillation of the investigational product (on the next day of surgery) (except instillation of non-steroidal anti-inflammatory ophthalmic solution at 3, 2, 1 and 0.5 hours before surgery)
* Patients with endogenous uveitis
* Patients planning to undergo surgery of the contralateral eye during the study period
* Patients with new intraocular bleeding after surgery
* Patients receiving gas or silicon oil in the vitreous body
* Patients with glaucoma or ocular hypertension (IOP on the next day of surgery ≥25 mmHg)
* Patients with superficial punctuate keratopathy or corneal ulcer
* Patients with any viral, bacterial or fungal keratoconjunctival disease
* Patients with allergy to any corticosteroid
* Patients requiring use of contact lens during the study period
* Women who were or might be pregnant, or lactating women
* Patients participating in another clinical study within 3 months before initiation of the present study
* Patients undergoing surgery under systemic anesthesia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2003-04; Study Completion 2003-07

PRIMARY OUTCOMES:
The variation from baseline in anterior chamber cell score on Day 14 (difference from baseline
score) was compared between the test and control groups.

SECONDARY OUTCOMES:
The variations from baseline in anterior chamber cell score on Days 3 and 7 were compared
between the test and control groups.
The numbers of patients with an anterior chamber cell score of 0 on Days 7 and 14 were
compared between the test and control groups.
The variations from baseline in anterior chamber flare score on Days 3, 7 and 14 were
The variations from baseline in total sign and symptom scores on Days 3, 7 and 14 were

CONTACTS AND LOCATIONS:
Overall Officials: Shigeaki Ohno, Study Chair — Professor, Department of Ophthalmology and Visual Science, Graduate School of Medicine, Hokkaido University